CLINICAL TRIAL: NCT04398082
Title: TRANslating Sleep Health Into QUaLity of Recovery (TRANQUiL) Study: A Multi-center Prospective Cohort Study of Sleep Health and Activity Measures Predicting Meaningful and Patient-centric Outcomes Following Non-cardiac Surgeries.
Brief Title: TRANslating Sleep Health Into QUaLity of Recovery (TRANQUiL) Study
Acronym: TRANQUiL
Status: Active, not recruiting | Type: Observational
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0044-B
Record Dates: First submitted 2019-10-24; First posted 2020-05-21 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disorder; Sleep Disturbance
Keywords: sleep
MeSH Terms: conditions — Sleep Wake Disorders; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a novel observational study with the overarching aim of evaluating the association between poor sleep health and poor quality of recovery in a surgical setting. It hopes to assess and optimize the perioperative sleep health of patients so significant improvements in their quality of recovery and health outcomes may be achieved.

DETAILED DESCRIPTION:
Surgery and pain may cause sleep disturbances that affect both physical and mental well-being of patients. Sleep disturbance can cause an increased risk of confusion after surgery, increased pain needing some or more medication, untoward events (heart and breathing problems), delayed recovery and increased lengths of hospital stay.

Hospitalization interferes with sleep patterns, causing poor quality sleep due to noise, light, pain, medication administration and nursing checks. The circadian rhythm, which is the "body clock" is a 24-hour cycle that tells our bodies when to sleep and rise. This in turn helps in regulating many physiological processes in the body. Sleep disruption affects the body clock, thereby changing hormone levels that may be responsible for poor wound healing. This study aims to evaluate sleep problems before disruption post-operatively and also evaluate the relation between poor sleep health and quality of recovery utilizing sleep health measurements such as sleep quality, sleep timing, and sleep efficiency.

Objectives of the study:

1. To examine the associations between specific pre-operative sleep-health parameters, predicting poor sleep health, and patient-centered outcomes such as pain control, delirium, sleep-related quality of life, and quality of recovery scores in the peri-operative period.
2. To estimate the association between presence of intrinsic sleep disorders and patient centric outcomes such as pain control, delirium, sleep-related quality of life and quality of recovery scores in the post-operative period.
3. To validate a set of subjective and objective measures of various sleep health domains in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years).
2. ASA physical status I - IV.
3. Undergoing elective primary or revision lower limb joint replacement surgeries (such as total or partial hip or knee replacement).

Exclusion Criteria:

1. Patients undergoing emergency surgeries; cardiac, trauma, organ transplantation or organ retrieval, obstetric or intracranial neurosurgeries.
2. Pregnant or lactating patients.
3. Inability to wear study-related monitoring devices per instruction or provide informed consent limiting adherence to protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 260 patients will be recruited from the preoperative clinics at major academic centers: Women's College Hospital (WCH) - Coordinating center, Toronto Western Hospital (TWH) - University Health Network (UHN); and St. Michaels Hospital (SMH), Toronto, Ontario.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery-15 score at 48 hrs postoperatively | 48 hours postoperatively
  QoR-15 Score is a validated patient-reported outcome questionnaire that measures the quality of recovery after surgery and anesthesia. Aggregate changes in QoR-15 scores (e.g., mean and SD) will be reported.
The diagnostic accuracy of each of the actigraphy derived measures | 48 hours postoperatively
  The diagnostic accuracy of each of the actigraphy derived measures with reference to the standard test will be calculated using the Receiver Operating Characteristic (ROC) curve, Sensitivity, Specificity, Positive predictive value (PPV), Negative predictive value (NPV), Positive Likelihood ratio, Negative Likelihood ratios, and Diagnostic Odds Ratio (DOR).

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) Scores | 3 months postoperatively
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized sleep questionnaire for multiple populations. It has seven component scores and a composite score to assess sleep health and daytime dysfunction in the past month.
Consensus Sleep Diary (CSD) Scores | 7 days prior surgery, 7 days, and 3 months postoperatively
  The Consensus Sleep Diary (CSD) is a standardized, prospective tool for tracking nightly subjective sleep.
Functional Outcomes in Sleep Questionnaire (FOSQ) | 7 days prior surgery and 3 months postoperatively
  The short-form FOSQ-10 scale has good psychometric properties with increased usability. It is a disease-specific instrument designed to assess the sleep-related quality of life measures.
Hospital Anxiety and Depression Scale (HADS) | Baseline and 3 months postoperatively
  The HADS is a very brief, easy to use screening measure comprising of 14 items measuring cognitive and emotional aspects of anxiety and depression. It has good psychometric properties for medical patients.
Fluid Intake and Output | 48 hours
  Postoperative assessment of the fluid intake and output.
Visual analogue pain scores (VAS) | 48 hours
  The VAS is a simple way for patients to rate the intensity of their pain. This pain scale shows a 10-centimeter line printed on a piece of paper, with anchors at either end and marked from 0-10. At one end is "no pain," and at the other end are "pain as bad as it could be" or "the worst imaginable pain."
Postoperative complications | 48 hours and 30 days
  Assessment of the severity of the postoperative complications
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Baseline and 3 months postoperatively
  The WOMAC questionnaire assesses the three dimensions of pain, disability and joint stiffness in knee and hip osteoarthritis using a battery of 24 questions in 5-point Likert, 100mm Visual Analogue and 11-box Numerical Rating Scale formats. It is a valid, reliable and responsive measure of outcome, and has been used in diverse clinical and interventional environments.
Epworth Sleepiness Scale (ESS) | Baseline and 3 months postoperatively
  The ESS is self-administered where the subjects are asked to rate on 0-3 scales how likely they would be to doze off or fall asleep in the eight situations. A summary score is generated where total score of >10 indicates excessive daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, MSc, Principal Investigator — Women's College Hospital and Toronto Western Hospital, University Health Network
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hospital (University Health Network), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided